CLINICAL TRIAL: NCT03821272
Title: A Phase I/II Clinical Trial of PepCan in Head and Neck Cancer Patients in Remission to Reduce Recurrence Regardless of HPV Status
Brief Title: A Phase I/II Clinical Trial of PepCan in Head and Neck Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 217672
Record Dates: First submitted 2019-01-23; First posted 2019-01-29 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer
Keywords: Squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: PepCan or placebo randomized at a 3:1 ratio in a double-blinded design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PepCan (Experimental): Four injections (one every 3 weeks) of PepCan, then three injections (one every 3 months) of PepCan for a total of 7 injections.
  Interventions: Biological: PepCan
- Placebo (Placebo Comparator): Four injections (one every 3 weeks) of placebo, then three injections (one every 3 months) of placebo for a total of 7 injections.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PepCan — 50 μg peptide + 0.3mL Candin® per dose administered intradermally in the extremities
  Other Names: HPV 16 E6 peptides combined with Candin®; PepCan Vaccine Regime
  Arms: PepCan
Biological: Placebo — 0.9% Saline solution per dose administered intradermally in the extremities
  Other Names: Saline; Placebo Vaccine Regimen
  Arms: Placebo

SUMMARY:
This study has been designed to evaluate the safety and efficacy of giving seven injections of PepCan or placebo over approximately a 24-month period in subjects with head and neck cancers who achieved remission. PepCan may prove to be beneficial in treating many stages of HPV-related malignancies starting from infection to cancer. Safety, efficacy in terms of reduced cancer recurrence, immunological responses and profiles, and gut microbiome changes will be assessed.

DETAILED DESCRIPTION:
This is a Phase I/II study to evaluate the efficacy and safety of an HPV therapeutic vaccine called PepCan (HPV-16 E6 peptides) in adults over a two (2) year period. Each subject will be receiving a total of 7 injections of PepCan (50 µg per peptide dose) or placebo (saline) at a 3:1 ratio in a randomized double-blinded design. Subjects will receive one injection every 3 weeks until they receive 4 injections. Then, subjects will receive one injection every 3 months until they receive a total of 7 injections. Subjects will have 2 more visits approximately 6 months apart after the last injection. Immunological assessment by enzyme-linked immunospot (ELISPOT) assay will be made at 4 time points (Visits 1, 5, 8, and 9), and by fluorescent activated cell sorter analysis will be made at times points at Visits 1, 3, 5, 6, 7, 8, and 9. Oral wash samples and stool samples will be collected at the Screening Visit, Visit 5, Visit 7 and Visit 8 for microbiome diversity analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Male or female 18 years of age or older
3. Squamous cell carcinoma of the head and neck who have completed curative therapy (surgery and/or radiation and/or chemotherapy) therapy within the previous 120 days
4. Performance status of Eastern Cooperative Oncology Group (ECOG) 0-2
5. No Evidence of Disease (NED) based on clinical and/or radiographic evaluations
6. Vital Signs recorded

   1. Blood pressure (≤160/95 mm Hg acceptable)
   2. Heart rate (50-100 beats per min acceptable)
   3. Respiratory rate (≥ 12 ≤25 breaths per min acceptable)
   4. Temperature (≤100°F acceptable)
7. Blood work done at Screening Visit

   1. White count (≥3x109/L acceptable)
   2. Hemoglobin (≥ 7 g/dL acceptable)
8. Willing and able to comply with the requirements of the protocol

Exclusion Criteria:

1. Positive urine pregnancy test for women of childbearing potential
2. Being pregnant or attempting to be pregnant within the period of study participation
3. Women who are breast feeding or plan to breast feed within the period of study participation
4. Patients who are allergic to Candin® or yeast
5. History of severe asthma requiring emergency room visit or hospitalization within the past 5 years
6. Patients who have previously received PepCan
7. History of recurrence of squamous cell carcinoma of the head and neck
8. If in the opinion of the Principal Investigator or other Investigators, it is not in the best interest of the patient to enter or continue in this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar T Atiq, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PepCan | Placebo
Started | 12 | 5
Completed | 9 | 5
Not Completed | 3 | 0
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PepCan | Placebo | Total
Number analyzed (Participants) | 12 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.03 (8.30) | 59.34 (14.00) | 59.82 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 11 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 5 | 17
White blood cells [Mean (Standard Deviation); unit: 10^3 cells/μL] — White blood cell count in blood
  10^3 cells/μL | 5.20 (1.52) | 4.64 (1.70) | 5.03 (1.55)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] — Hemoglobin amount in blood
  g/dL | 11.94 (1.91) | 10.88 (1.43) | 11.63 (1.81)
Hematocrit [Mean (Standard Deviation); unit: %] — Hematocrit is an indication of the percentage of blood volume composed of red blood cells.
  % | 36.63 (5.73) | 32.96 (4.64) | 35.55 (5.56)
Body mass index [Mean (Standard Deviation); unit: kg/m2] — Body mass index is a measure of body fat based on weight divided by height squared.
  kg/m2 | 22.30 (3.82) | 21.86 (4.41) | 22.17 (3.87)
Human papillomavirus status [Count of Participants; unit: Participants]
  Positive | 0 | 0 | 0
  Negative | 0 | 1 | 1
  Unknown | 12 | 4 | 16
P16 [Count of Participants; unit: Participants] — P16 is a surrogate marker for human papillomavirus infection.
  Participants
    P16 positive | 4 | 3 | 7
    P16 negative | 5 | 0 | 5
    P16 unknown | 3 | 2 | 5
Human Papillomavirus/P16 [Count of Participants; unit: Participants] — Ratio of human papillomavirus to P16 status.
  Participants
    HPV/P16 positive | 4 | 3 | 7
    HPV/P16 negative | 5 | 1 | 6
    HPV/P16 unknown | 3 | 1 | 4
Tumor location [Count of Participants; unit: Participants]
  Site: Pharynx | 6 | 5 | 11
  Site: Larynx | 3 | 0 | 3
  Site: Oral | 3 | 0 | 3
TNM Staging, Tumor [Count of Participants; unit: Participants] — The TNM staging system is a widely-used system for staging different types of cancer. The T portion of TNM refers to the size and extent of the main, or primary, tumor.
  Here, the frequency of participants with a given T stage is what is reported here.
  Higher grades/stages (e.g., T4) indicate larger tumors or more invasion into surrounding tissues.
  Participants
    TNM Staging, Tumor: T1 | 3 | 0 | 3
    TNM Staging, Tumor: T2 | 2 | 4 | 6
    TNM Staging, Tumor: T3 | 3 | 1 | 4
    TNM Staging, Tumor: T4 | 4 | 0 | 4
TNM Staging, Lymph node [Number; unit: participants] — The TNM staging system is a widely-used system for staging different types of cancer. The N portion of TNM refers to the number of nearby lymph nodes that have cancer.
  Here, the frequency of participants with a given N stage is what is reported here.
  Higher grades (e.g., N3) indicate more spread to nearby lymph nodes.
  participants
    TNM Staging, Lymph node: N0 | 1 | 1 | 2
    TNM Staging, Lymph node: N1 | 1 | 2 | 3
    TNM Staging, Lymph node: N2 | 8 | 2 | 10
    TNM Staging, Lymph node: N3 | 2 | 0 | 2
TNM Staging, Metastasis: M0 [Number; unit: participants] — Metastasis portion of the TNM Staging system, which is a cancer staging system.
  The TNM staging system is a widely-used system for staging different types of cancer. The M portion of TNM refers to whether the cancer has metastasized, or spread from the primary tumor to other parts of the body.
  Here, the frequency of participants with a given M stage is what is reported here.
  MX means that the metastasis cannot be measured. M0 means the cancer has not spread to other parts of the body. M1 means the cancer has spread to other parts of the body.
  participants
    MX | 0 | 0 | 0
    M0 | 12 | 5 | 17
    M1 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events - Evaluate Safety of a 7-injection Regimen of PepCan.
Description: To evaluate the safety of a 7-injection regimen of PepCan, adverse events will be captured and assessed per NCI CTCAE Version 5.0 whether they are treatment-related or not by a physician.
Time Frame: 2 years
Population: Participants with side effects occurring with 5% or more injections.
Measure: Number; unit: adverse event
Arm/Group | PepCan | Placebo
Number analyzed (Participants) | 12 | 5
adverse event
  General Disorders and Site Administration Conditions: Injection site reaction | 23 | 0
  General Disorders and Site Administration Conditions: Fatigue | 0 | 1
  Immune System Disorders : Allergic reaction | 2 | 0
  Injury, Poisoning and Procedural Complications : Vaccination complication | 4 | 1
  Metabolism and Nutrition Disorders: Hypokalemia | 1 | 0
  Nervous System Disorders : Dizziness | 1 | 0
  Nervous System Disorders : Headache | 2 | 0
  Skin and Subcutaneous Tissue Disorders : Pruritus | 1 | 0

2. Secondary Outcome: Cancer Recurrence Rate - Efficacy of a 7-injection Regimen of PepCan
Description: To evaluate the efficacy, cancer recurrence rates will be compared between the PepCan and placebo arms. Patients with a "non-recurrence" status are defined as responders. Patients with a "recurrence" status are defined as non-responders.
Time Frame: Study completion, approximately 24 months after enrollment
Population: Patients who screen-failed or were considered ineligible were excluded from the ITT analysis and PP analysis..
Measure: Count of Participants; unit: Participants
Arm/Group | PepCan | Placebo
Number analyzed (Participants) | 12 | 5
Participants
  Non-recurrence | 5 | 4
  Recurrence | 4 | 1
  Withdrawn | 2 | 0
  Ineligible | 1 | 0

3. Secondary Outcome: Efficacy Analysis (Intention to Treat) - PepCan
Description: Patients with a "non-recurrence" status are defined as responders. Patients with a "recurrence" status are defined as non-responders. The Intention-to-Treat outcome is based on the worst-case scenario and considers those who withdrew as non-responders. Patients who screen-failed or were considered ineligible were excluded from the ITT analysis.
Time Frame: Study completion, approximately 24 months after enrollment
Population: Patients who screen-failed or were considered ineligible were excluded from the ITT analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PepCan
Number analyzed (Participants) | 12
Participants
  Responder | 5
  Non-responder | 6
  Unknown | 1
Statistical Analysis 1: Comparison: PepCan; Test type: Superiority; p = 0.31, Fisher Exact; non-recurrence rate = 0.45, 95% CI 2-sided [0.17 to 0.77]

4. Secondary Outcome: Efficacy Analysis (Intention to Treat) - Placebo
Description: as for outcome 3
Time Frame: Study completion, approximately 24 months after enrollment
Population: Patients who screen-failed or were considered ineligible were excluded from the ITT analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 5
Participants
  Responder | 4
  Non-responder | 1
  Unknown | 0
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.31, Fisher Exact; non-recurrence rate = 0.80, 95% CI 2-sided [0.28 to 0.99]

5. Secondary Outcome: Efficacy Analysis (Per Protocol) - PepCan
Description: The Per Protocol outcome includes subjects who completed the study either by completing Visit 9 or having had recurrences. Patients who screen-failed, withdrew, or were considered ineligible (after randomization) are excluded from the PP analysis.
Time Frame: Study completion, approximately 24 months after enrollment
Population: Patients who screen-failed, withdrew, or were considered ineligible (after randomization) are excluded from the PP analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PepCan
Number analyzed (Participants) | 12
Participants
  Responder | 5
  Non-responder | 4
  Unknown | 3
Statistical Analysis 1: Comparison: PepCan; Test type: Superiority; p = 0.58, Fisher Exact; non-recurrence rate = 0.56, 95% CI 2-sided [0.21 to 0.86]

6. Secondary Outcome: Efficacy Analysis (Per Protocol) - Placebo
Description: as for outcome 5
Time Frame: Study completion, approximately 24 months after enrollment
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 5
Participants
  Responder | 4
  Non-responder | 1
  Unknown | 0
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.58, Fisher Exact; non-recurrence rate = 0.80, 95% CI 2-sided [0.28 to 0.99]

ADVERSE EVENTS:
Time Frame: Approximately 24 months
Description: Not based on a different definition of adverse event and/or serious adverse event than the Adverse Events definition on clinicaltrials.gov
Arm/Group | PepCan | Placebo
All-Cause Mortality (participants affected / at risk) | 1/12 | 0/5
Serious Adverse Events (participants affected / at risk) | 5/12 | 2/5
Other Adverse Events (participants affected / at risk) | 12/12 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PepCan (N=12) | Placebo (N=5)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 (3) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PepCan (N=12) | Placebo (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 6 (7) | 0 (0)
Allergic reaction (Immune system disorders) | 3 (3) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 10 (18) | 5 (12)
Anorexia (Metabolism and nutrition disorders) | 5 (6) | 2 (4)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood antidiuretic hormone abnormal (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (3) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Creatinine increased (Investigations) | 3 (3) | 2 (3)
Depression (Psychiatric disorders) | 4 (4) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 10 (17) | 5 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 7 (10) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 9 (15) | 4 (9)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Edema face (General disorders) | 2 (2) | 1 (2)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Facial pain (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 8 (8) | 4 (5)
Fever (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 (8) | 2 (7)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 5 (5) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (9) | 2 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 7 (8) | 3 (5)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (5) | 5 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (14) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 6 (10) | 5 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 5 (8) | 3 (5)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 10 (23) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Investigations - Other, specify (Investigations) | 9 (33) | 3 (13)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 11 (34) | 5 (19)
Malaise (General disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (5)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (3) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (4) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (2) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (5)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 (4) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 4 (5) | 3 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (4) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Weight loss (Investigations) | 5 (9) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 4 (10) | 3 (10)
Neck edema (General disorders) | 3 (3) | 1 (1)
Bone infection (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scleral disorder (Eye disorders) | 1 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT03821272/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT03821272/ICF_000.pdf